CLINICAL TRIAL: NCT07309874
Title: Effect of Ultrasound-Guided Dry Needling Targeting Rectus Capitus Posterior Major on Individuals With Headaches
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Texas Tech University Health Sciences Center (Other)
Collaborators: Texas Woman's University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-FY2026-36; No funding number available (Other Grant/Funding Number: Texas Society for Advancement of Health Professions Research and Innovative Practice Grant Award)
Record Dates: First submitted 2025-11-20; First posted 2025-12-30 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Headache Disorders, Primary; Headache, Cervicogenic
Keywords: Headache; cervical spine; suboccipital muscles; needle placement
MeSH Terms: conditions — Headache Disorders, Primary; Post-Traumatic Headache; Headache | interventions — Dry Needling

STUDY DESIGN:
Intervention Model Description: Each subject will receive two separate dry needle insertions targeting the rectus capitus posterior major. Method 1 will be 30 degrees (relative to the frontal plane) insertion angle toward the occiput. Method 2 will be 45 degrees (relative to the frontal plane) insertion angle toward the occiput.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dry needling (Experimental)
  Interventions: Other: Dry needling

INTERVENTIONS:
Other: Dry needling — Each subject will receive two separate dry needle insertions targeting the rectus capitus posterior major. Method 1 will be 30 degrees (relative to the frontal plane) insertion angle toward the occiput. Method 2 will be 45 degrees (relative to the frontal plane) insertion angle toward the occiput.

SUMMARY:
Headaches such as tension-type, migraine, and cervicogenic (neck-related) headaches are among the most common and disabling conditions worldwide. and are often associated with tight or sensitive muscles at the base of the skull, which can contribute to headaches. Dry needling involves inserting a very thin, sterile needle into tight muscle areas known as trigger points to relieve pain and muscle tension. When applied to the deep neck muscles, including those beneath the skull, dry needling may reduce headache symptoms. The suboccipital region contains important structures such as the vertebral artery, greater occipital nerve, and spinal cord, which requires precise needle placement to maintain safety. Many needling techniques used in this region have not been validated for accuracy or safety in living subjects. This study will use real-time ultrasound imaging to guide dry needling of the rectus capitis posterior major muscle and directly visualize nearby structures to minimize risk.

The main goals of this research are to examine the effects of a single session of ultrasound-guided dry needling on headache symptoms and to confirm the safety, accuracy, and consistency of the proposed needling technique using ultrasound imaging.

DETAILED DESCRIPTION:
RESEARCH DESIGN: Prospective, single-arm, repeated-measures interventional study with secondary observational ultrasound validation of two insertion angles and intra-rater test-retest reliability of ultrasound assessments at ~6 months.

PROCEDURE: Each participant will complete one study visit lasting approximately 60 minutes. During each data collection session:

1. Screening: Participants will undergo screening for inclusion and exclusion criteria.

   o Eligible participants will then complete: A Numeric Pain Rating Scale (NPRS) of their headache pain on a scale from 0 to 10 (0 = no pain; 10 = worse pain) including: Current rating; Best rating; Worst rating in the past 6 months; Complete the Headache Disability Index (HDI)
2. Positioning: Participants will be positioned prone on a treatment table with cervical spine alignment monitored using an inclinometer to ensure cervical lordosis is under 10°.
3. Landmark Identification & Needle Insertion:

   * Landmark Identification: The PI will palpate and mark two bony landmarks in the upper neck including: 1. The C2 Spinous process, a distinct bone that can be felt at the top of the spine below the skull, and 2. The C1 Transverse process, a bony ridge located just below and slightly to the side of the base of the skull at ~45-degree angle from the ear. (These landmarks will help determine the correct location for the needle insertion.)
   * Needle Insertion: Sterile, 0.25 gauge/diameter, 40 mm needles will be used. A new needle will be used for each individual needle insertion before being discarded in a sharps container. The needle will be inserted just below the base of the skull, slightly off the center line of the neck. Each participant will have two separate needle insertions during the single data collection visit. Two dry needle insertion techniques will be performed in a randomized order: Method 1: 30° (relative to the frontal plane) insertion angle toward the occiput, and Method 2: 45° (relative to the frontal plane) insertion angle toward the occiput.
   * Needle Target: The target of the needle is a deep muscle (Rectus Capitus Posterior Major) that attaches to the base of the skull (occiput). For both methods, the needle will be advanced until bony contact is achieved, and then slightly pulled in/out within the muscle to visualize needle placement on ultrasound
   * Randomization of technique order (Method 1 vs. Method 2) will be generated using the list randomizer from https://www.random.org/lists/
4. Ultrasound Imaging: An investigator will use a Sonosite PX ultrasound device to capture still images and 3-second video clips of needle placement relative to the RCPMaj and surrounding anatomy. Participants may be asked to laterally deviate their eyes to assist in muscle visualization.
5. Data Collection: Investigators will record whether a bony backdrop was felt, if the needle reached the RCPMaj, and the length of unused needle remaining outside the skin as well as if the needle pierce through the vertebral artery.

IMMEDIATE POST-PROCEDURE: Participants will be asked to rate their current level of pain immediately following the intervention on the NPRS from 0 to 10 (0 = no pain; 10 = worse pain)

POST-PROCEDURE FOLLOW UP VISIT: 24-48 hours following data collection, participants will be asked to complete the following via a secure, anonymous online survey link to the electronic platform Qualtrics®. Participants will be sent an email with the secure survey link and reminder of their unique study ID. Participants will only use their unique assigned study ID. No identifying information (name, email address, or IP address) will be collected in Qualtrics® survey responses. Participants will report: 1) Post-needling soreness (Yes/No), 2) NRPS including Current rating, Best rating and Worst rating in the last 24-48 hours, and 3) Headache Disability Index

ELIGIBILITY:
Inclusion Criteria:

* Reports of a headache within the last 6 months (no minimum or maximum frequency or duration)
* Current reports of headache
* Tenderness to palpation of suboccipital muscles with Numeric Pain Rating Scale score ≥ 2/10
* No history of cervical spine surgery or neurological disorders

Exclusion Criteria:

* History of cervical spine trauma or surgery
* Diagnosed bleeding disorder
* Currently using anticoagulant medications
* Currently using anti-platelet medications
* Diagnosed systemic joint diseases such as rheumatoid arthritis
* Active infection
* Diabetes
* Cancer
* Fibromyalgia
* Cervical radiculopathy
* Inability to tolerate prone positioning for the duration of the procedure.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Post-needling soreness | 24-48 hours post-data collection
  Subjective outcome measures:
  • Post-data collection reports of post-needling soreness (Dichotomous report: Yes or No)
Numeric Pain Rating Scale | Baseline immediately pre-data collection and then again 24-48 hours post-data collection
  Numeric Pain Rating Scale (0 = no pain; 10 = worst pain): Pre-data collection will include Current rating, Best rating in past 6 months, and Worst rating in past 6 months. Post-data collection will include Current rating, Best rating in past 24-48 hours, and Worst rating in past 24-48 hours
Headache Disability Index | Baseline immediately pre-data collection and then again 24-48 hours post-data collection
  Headache Disability Index: Scores range from 0 to 100. A total score of 10-28 is considered mild disability. A total score of 30-48 is considered moderate disability. A total score of 50-68 is severe disability. A total score of 72-100 is considered complete disability. Participants will complete the Headache Disability Index immediately pre-data collection and then 24-48 hours post-data collection

SECONDARY OUTCOMES:
Frequency of needle placement reaching a bony structure | Baseline
  For each needle insertion, a dichotomous decision (Yes vs. No) will be made via ultrasound imaging if the needle reached the occiput (bony structure)
Frequency of successful needle placement into the Rectus Capitus Posterior Major | Baseline
  For each needle insertion, a dichotomous decision (Yes vs. No) will be made via ultrasound imaging if the needle reached the Rectus Capitus Posterior Major
Length of unused needle at the point of bony contact | Baseline
  For each needle insertion, the length of needle remaining outside the skin will be measured in millimeters for each time the needle reaches the occiput (bony contact)

OTHER OUTCOMES:
Intra-rater Reliability: Frequency of needle placement reaching a bony structure | Baseline during primary data collection and then again 6 months post-data collection
  Intra-rater reliability (Cohen's kappa) will be calculated for identification of needle placement at time 0 and 6-month follow-up review. Investigators will assess secondary outcomes of frequency of needle placement reaching a bony structure at time 0 (baseline) and then again at 6 months post-data collection. The 6 month post-data collection decisions will be made from a 10 second video clip taken during primary data collection
Intra-rater Reliability: Frequency of Needle Placement into Rectus Capitus Posterior Major | Baseline during primary data collection and then again 6 months post-data collection
  Intra-rater reliability (Cohen's kappa) will be calculated for identification of needle placement at time 0 and 6-month follow-up review. Investigators will assess secondary outcomes of frequency of successful needle placement into the Rectus Capitus Posterior Major at time 0 (baseline) and then again at 6 months post-data collection. The 6 month post-data collection decisions will be made from a 10 second video clip taken during primary data collection

CONTACTS AND LOCATIONS:
Overall Officials: Gary A Kearns, PT, ScD, Principal Investigator — Texas Tech University Health Sciences Center

IPD SHARING:
Plan to Share IPD: No
There is no need to share IPD with other investigators. Once completed, there will be no need to access any IPD in the future.

REFERENCES:
- [Background] Kearns GA, Lierly M, Gilbert KK, Dommerholt J. Guidelines to minimize risk when dry needling the rectus capitus posterior major muscle. Musculoskelet Sci Pract. 2025 Apr;76:103260. doi: 10.1016/j.msksp.2025.103260. Epub 2025 Jan 10. PMID 39823665
- [Background] Kearns GA, Hooper TL, Brismee JM, Allen B, Lierly M, Gilbert KK, Pendergrass TJ, Edwards D. Influence of clinical experience on accuracy and safety of obliquus capitus inferior dry needling in unembalmed cadavers. Physiother Theory Pract. 2022 Dec;38(12):2052-2061. doi: 10.1080/09593985.2021.1901326. Epub 2021 Mar 15. PMID 33719823
- [Background] Kearns G, Fernandez-De-Las-Penas C, Brismee JM, Gan J, Doidge J. New perspectives on dry needling following a medical model: are we screening our patients sufficiently? J Man Manip Ther. 2019 Jul;27(3):172-179. doi: 10.1080/10669817.2019.1567011. Epub 2019 Jan 19. PMID 30935332
- [Background] GBD 2016 Headache Collaborators. Global, regional, and national burden of migraine and tension-type headache, 1990-2016: a systematic analysis for the Global Burden of Disease Study 2016. Lancet Neurol. 2018 Nov;17(11):954-976. doi: 10.1016/S1474-4422(18)30322-3. PMID 30353868
- [Background] Stovner LJ, Hagen K, Linde M, Steiner TJ. The global prevalence of headache: an update, with analysis of the influences of methodological factors on prevalence estimates. J Headache Pain. 2022 Apr 12;23(1):34. doi: 10.1186/s10194-022-01402-2. PMID 35410119
- [Background] Jung A, Carvalho GF, Szikszay TM, Pawlowsky V, Gabler T, Luedtke K. Physical Therapist Interventions to Reduce Headache Intensity, Frequency, and Duration in Patients With Cervicogenic Headache: A Systematic Review and Network Meta-Analysis. Phys Ther. 2024 Feb 1;104(2):pzad154. doi: 10.1093/ptj/pzad154. PMID 37941472
- [Background] Pourahmadi M, Dommerholt J, Fernandez-de-Las-Penas C, Koes BW, Mohseni-Bandpei MA, Mansournia MA, Delavari S, Keshtkar A, Bahramian M. Dry Needling for the Treatment of Tension-Type, Cervicogenic, or Migraine Headaches: A Systematic Review and Meta-Analysis. Phys Ther. 2021 May 4;101(5):pzab068. doi: 10.1093/ptj/pzab068. PMID 33609358
- [Background] Navarro-Santana MJ, Sanchez-Infante J, Fernandez-de-Las-Penas C, Cleland JA, Martin-Casas P, Plaza-Manzano G. Effectiveness of Dry Needling for Myofascial Trigger Points Associated with Neck Pain Symptoms: An Updated Systematic Review and Meta-Analysis. J Clin Med. 2020 Oct 14;9(10):3300. doi: 10.3390/jcm9103300. PMID 33066556
- [Background] Chys M, De Meulemeester K, De Greef I, Murillo C, Kindt W, Kouzouz Y, Lescroart B, Cagnie B. Clinical Effectiveness of Dry Needling in Patients with Musculoskeletal Pain-An Umbrella Review. J Clin Med. 2023 Feb 2;12(3):1205. doi: 10.3390/jcm12031205. PMID 36769852